CLINICAL TRIAL: NCT04709926
Title: Paramedic Experiences and Perceptions of Training for Participation in Research: the PREPARE Study
Acronym: PREPARE
Status: Withdrawn | Type: Observational
Why Stopped: Capacity issues within team after pandemic & unable to progress with the study
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00686
Record Dates: First submitted 2020-01-16; First posted 2021-01-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Staff Attitude
Keywords: PRESTO study; Research training; Paramedics
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paramedics that were eligible to take part in the PRESTO study: Paramedics that are employed by one of the four Ambulance Services involved in the PRESTO study and were eligible to complete the training provided by Manchester University NHS Foundation Trust to take part in the PRESTO study.
  Interventions: Other: Survey; Other: Interview (optional)

INTERVENTIONS:
Other: Survey — Paramedics will complete a 5 minute survey that is asking for their opinions on why they did or did not take part in the PRESTO training package and also why they think paramedics might not engage with research training in general.
Other: Interview (optional) — Paramedics will also be given the option to participate in a 1hr interview to explore the questions asked in the survey in more detail.

SUMMARY:
The investigators are currently conducting a research study, called PRESTO, in the pre-hospital environment where the investigators are asking paramedics to talk to patients about participating in the research study, interpret a heart tracing (or ECG), take a blood sample and record some study specific information. Apart from ECG interpretation, these are activities that the paramedics would not normally do and so the investigators had to provide training in order to ensure that these activities were carried out to the same standard across the four ambulance services that were involved, all of who have different working practices.

In order to do this, the investigators provided a training package based around four subject areas - blood sample collection, heart tracing interpretation, background to the study and the importance of conducting the study activities to a high standard (called Research Fundamentals). These were presented to the paramedics either as online training or in a face-to-face session. There has been a mixed response to both the uptake in training across the four ambulance services and the engagement from paramedics in following PRESTO with a potential participant.

As more research is being done in the pre-hospital environment the investigators feel that it would be beneficial to try to find out why paramedics may or may not have taken part in the PRESTO training. To do this the investigators will be sending out a survey to each of the four ambulance services which will contain questions around whether the paramedics thought the training package for PRESTO was suitable, whether the paramedics felt confident following PRESTO with a potential participant after the training and what the paramedics think the main barriers are to participating in research. Up to 30 paramedics will also be approached to participate in an interview, which will explore these ideas further.

This should allow the investigators to identify potential barriers that prevent paramedics from taking part in training for research studies. It should also allow the investigators to offer insight to future researchers about the type of training that should be provided for paramedics for a research study and how it should be delivered.

ELIGIBILITY:
Inclusion Criteria:

* Staff that are employed by one of the four ambulance services involved in the PRESTO study

Exclusion Criteria:

* Staff that are not employed by one of the four ambulance services involved in the PRESTO study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Staff employed by one of the four ambulance services that were involved in the PRESTO study Paramedics that either did or did not complete the PRESTO training package are eligible to take part as we would like to get opinions from both groups.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Paramedic views on research training via survey | For the study duration, an average of 5 months
  Survey will be used to collect answers on paramedics' views of training for research studies
Paramedic views on research training via interview (optional) | For the study duration, an average of 5 months
  Interview will be used to collect answers on paramedics' views of training for research studies

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No